CLINICAL TRIAL: NCT03319394
Title: The First Twenty Exercise Training Program and Fire Academy Recruits' Fitness and Health
Brief Title: The First 20 Fire Academy Recruits Exercise Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: National Development and Research Institutes, Inc. (Other)
Responsible Party: Principal Investigator, Katie M. Heinrich, Associate Professor, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8063
Record Dates: First submitted 2017-10-13; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Physical Fitness
Keywords: Firefighters; Exercise Training; Resistance Training; Exercise Test; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study statistician did not know which condition participants were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The First Twenty (Experimental): TF20 group completed a structured exercise program. Once a week a trained firefighter with current CPR and First Aid certifications met with the group to assess progress and answer questions about the workouts or the program. The rest of the time, the participants completed the workouts on their own time. Workouts contained a combination of aerobic (e.g., running, rowing, jumping), body weight (e.g., air squats, pushups, situps), and weight lifting (e.g., presses, back squats, lunges) exercises with workouts designed to use equipment available in an exercise/gym facility (e.g., weight racks, benches). Sixty-minute TF20 sessions included a warm-up, workout and cool down. All sessions were able to be logged online in TF20 program.
  Interventions: Behavioral: The First Twenty
- Comparison (Active Comparator): The Comparison Group followed and documented their regular workout routine for 14 weeks. Once a week, a trained firefighter with current CPR and First Aid certifications met with the group to discuss questions. Participants were able to choose when to complete their workouts.
  Interventions: Behavioral: Comparison

INTERVENTIONS:
Behavioral: The First Twenty — The First Twenty workouts were part of an online training program that provided resistance and endurance exercises, nutritional information, and mental performance guidance. The intervention, created by firefighters for firefighters, was a 10-week periodized program with workouts increasing in frequency and intensity each week.
  Arms: The First Twenty
Behavioral: Comparison — Documentation of having previously taken or concurrent enrollment in a 1 credit hour fitness class offered through the community college. HPER 240, Lifetime Fitness, introduced the student to basic fitness principles, physical activity and the relationship to a healthy lifestyle. The course was graded based on an initial assessment/orientation and participation; the student was required to log hours at the community college gym. This course was waived at the discretion of the Fire Academy Director if the student proved they had an active gym membership at a local gym facility.
  Arms: Comparison

SUMMARY:
"The First Twenty (TF20) Exercise Training Program and Fire Academy Recruits' Fitness and Health" was thesis research completed in the Functional Intensity Training Laboratory (FIT Lab) at Kansas State University. The purpose was to assess the performance outcomes, acceptability, feasibility, and preliminary efficacy of an innovative 14-week Firefighter Fitness and Wellness Program. This study explored if TF20 program was a valid preparatory program for fire academy recruits training for the physical job of a firefighter compared to standard care of taking a college fitness class. It was hypothesized that TF20 group would see greater fitness improvements than the comparison group, the training program would be acceptable and feasible, and that TF20 group would report higher levels of group cohesion.

DETAILED DESCRIPTION:
The First Twenty (TF20) is an innovative computer based firefighter training program that provides foundational educational principles around firefighter physical fitness, mental wellness, and nutrition and is much more cost effective than other fitness program options. The current Fire Academy at Johnson County Community College (JCCC) does little to address the physical fitness of its firefighter recruits other than the physical skills taught in class. The recruits are required to either have previously taken or be concurrently enrolled in a 1 credit hour fitness class offered through the community college. HPER 240, Lifetime Fitness, introduces the student to basic fitness principles, physical activity and the relationship to a healthy lifestyle. The course is graded based on an initial assessment/orientation and participation; the student must log so many hours at the JCCC Gym (JCCC, 2015). This course may be waived at the discretion of the Fire Academy Director if the student can prove they have an active gym membership at a local gym facility. The recruits participate in highly physically demanding tasks as they learn the job of a firefighter. Part of the class is spent indoors for lecture. The remainder of the class is spent on the drill ground learning basic firefighter skills such as donning bunker gear (personal protective equipment) and self-contained breathing apparatus (SCBA), navigating through dark search quarters, searching and removing a victim in a fire room, climbing ladders, cutting ventilation holes on flat and pitched roofs, and fighting live fire in a propane burn facility. The recruits are also required to take the Candidate Physical Ability Test (CPAT) during the Fire Academy. The CPAT is a timed physical ability test designed to assess the fitness of firefighter candidates and is used as a screening tool for hiring new firefighters. In addition to completing the current requirements for the Fire Academy, this study included a baseline assessment, 14- weeks of group exercise training, and a post-test assessment. Fire Academy recruits were required to have taken or be concurrently enrolled in a one credit hour gym class; this study took the place of that one credit hour physical requirement. Participants were randomly assigned to one of two exercise groups: TF20 or the Comparison Group (CG). TF20 group exercised five days per week for 14 weeks, similar to the requirements of the Lifetime Fitness (HPER 240) course; the Comparison Group were asked to continue their current exercise regimen (ie: HPER 240 course). Travel workout options were available for TF20 group. It was hypothesized that TF20 group would see greater fitness improvements than the comparison group, TF20 group would find the training program acceptable and feasible, and TF20 group would report higher levels of group cohesion than the comparison/control group.

ELIGIBILITY:
Inclusion Criteria:

* Accepted for admission into spring 2016 Johnson County Community College Fire Academy; did not answer "YES" to any of the PAR-Q questions.

Exclusion Criteria:

* Answering "YES" to any of the PAR-Q questions will require physician's clearance for participation in the study; known cardiovascular, metabolic, or respiratory disease, or having an internal pacemaker are all exclusionary criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2016-05-16 (Actual); Study Completion 2016-05-16 (Actual)

PRIMARY OUTCOMES:
Change Candidate Physical Ability Test Time | Week 0 and Week 11
  The CPAT consists of eight separate events. This test is a sequence of events that requires the candidate to progress along a predetermined path from event to event in a continuous manner. This is a pass/fail test based on a maximum total time of 10 minutes and 20 seconds.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) | Week 0 and Week 11
  Measured height in meters and measured weight in kilograms were used to calculate BMI as kg/m2
Change in Body Composition | Week 0 and Week 11
  A Tanita TBF-300 scale was used to measure changes in body fat percentage, fat mass, and fat free mass.
Change in Post Exercise Heart Rate | Week 0 and Week 11
  Heart Rate in beats per minute was assessed via a heart rate monitor immediately post-exercise
Change in Blood Pressure | Week 0 and Week 11
  An Omron BP785 10 series monitor will be used to assess blood pressure after the participant has been seated comfortably for at least 5 minutes.
Change in Estimated VO2Max | Week 0 and Week 11
  Sub-Maximal Graded Exercise Test using a StairMaster 7000pt
Change in Hand Grip Strength | Week 0 and Week 11
  A Hand Grip Dynamometer will be used to assess hand grip strength in kg
Change in Vertical Jump Height | Week 0 and Week 11
  A Vertec vertical jump tester will be used to measure jump height in cm
Change in Push-ups | Week 0 and Week 11
  Participants will complete as many push-ups repetitions as possible in 2 minutes
Change in Curl-ups | Week 0 and Week 11
  Participants will complete the American College of Sports Medicine curl-up 12-inch test
Change in Agility | Week 0 and Week 11
  Participants will complete the Agility T-Test
Change in Flexibility | Week 0 and Week 11
  Participants will complete the sit-and-reach test using a Flexometer

CONTACTS AND LOCATIONS:
Overall Officials: Katie M Heinrich, PhD, Principal Investigator — Kansas State University
Locations (1):
- Kansas State University, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hollerbach BS, Jahnke SA, Poston WSC, Harms CA, Heinrich KM. Examining a novel firefighter exercise training program on simulated fire ground test performance, cardiorespiratory endurance, and strength: a pilot investigation. J Occup Med Toxicol. 2019 Apr 23;14:12. doi: 10.1186/s12995-019-0232-2. eCollection 2019. PMID 31049072